CLINICAL TRIAL: NCT01688713
Title: Phase II Trial of Double Dose of Icotinib in Treating Brain Metastases From Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH-LCBM-1202
Record Dates: First submitted 2012-08-27; First posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Brain Metastases; Non-small Cell Lung Cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib,Brain metastases (Experimental)
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — The patients will receive Icotinib in doses of 250mg thrice per day until disease progression or undue toxicity.

SUMMARY:
Brain metastases, a common complication,occur in 25-40% of patients with non-small cell lung cancer (NSCLC). Whole-brain radiation therapy(WBRT) and Stereotactic Radiosurgery (SRS) are important approaches to the treatment of brain metastases from NSCLC. Known to us, epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) can pass through the blood-brain barrier and show promising antitumor activity against brain metastases from NSCLC, especially for EGFR mutation patients. However, due to the lower concentration of tyrosine kinase inhibitors (TKIs) in the cerebrospinal fluid and its inevitable emergence of drug resistance, brain metastases will be refractory or resistant to standard-dose EGFR inhibitors. Icotinib is one agent of EGFR-TKIs. The previous studies have shown that the Icotinib conventional dose (125mg, TID) is far from reached its maximum tolerable dose. It is a challenge whether the further dose escalation of Icotinib will enhance its concentration in cerebrospinal fluid and thereby improve its therapeutic effect. Here the investigators examine the therapeutic effect and side-effect of double dose of Icitinib in treating patients with brain metastases from NSCLC who have suffered from the failure of conventional dose treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologic diagnosis of NSCLC
* Patients with disease progression after local treatment(WBRT and/or SRS) combined with Icotinib treatment.
* Patients with EGFR mutation or the lesions that remains stable for more than 3 months after local treatment(WBRT and/or SRS) combined with Icotinib treatment.
* ECOG performance status 0-2
* Doctors consider the patients will not benefit from local treatment(WBRT and/or SRS)
* Expected survival of greater than 3 months
* Age: 18-75 years
* The patients with key organs maintenance of basic function: Hemoglobin ≥ 9g/dL, White Blood Cell ≥ 3×109/L, Neutrophil count ≥ 1.5×109/L, platelets ≥ 80×109/L, total bilirubin < 1.5 times of the upper normal values, Alanine transaminase (ALT) and aspartate transaminase (AST) < 2.5 of the upper normal values, the serum creatinine < 1.5 times of the upper normal values
* Signed informed consent document on file.

Exclusion Criteria:

* Brain metastasis without local treatment before
* Patients without the treatment of Icotinib before or the therapeutic time less than 3 months
* More than 3 extracranial organs have metastatic lesions
* The patient with other type malignant tumors before
* The patient with fertility capacity, but without contraceptive application

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-02 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (intracranial lesions) | 2 years

SECONDARY OUTCOMES:
Partial response rate of intracranial lesions | 2 years
Partial response rate of extracranial lesion | 2 years
Overall survival | 3 years
Health-related quality of life quality | 2 years
number of adverse events such as skin rash,diarrhea ,abnormal liver function and so on | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Mao, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China